# Full study protocol and statistical analysis plan

## Official Title of the study:

Soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin levels in women with premature ovarian insufficiency

### Date of the document:

November 2020.

#### Contents:

- 1. Participant Flow
- 2. Baseline Characteristics
- 3. Outcome Measures
- 4.Endpoints of the study
- 5.Limitations and Strengths
- 6. Certain Agreements
- 7. Results Point of Contact

#### 1. Participant Flow

#### Recruitment Details

This will be an observational prospective cohort study conducted at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between November 2020 and April 2021. We will be recruited 45 subjects with idiopathic POI, and 45 healthy patients were selected for the control group. All patients will be given their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2020/320). The study strictly will be adhered to the principles of the Declaration of Helsinki.

#### Pre-assignment Details

The authors first will be assessed the recruited people to ensure meeting the inclusion and exclusion criteria. The inclusion criteria will be made according to the official documents.

#### Arm/Group Information \*

There are two groups in the study.

#### Arm/Group Title \*

Premature ovarian insufficiency group

Control group

#### 2. Baseline Characteristics

Power analysis could not be performed since there was no research on POI with these three markers in the literature. Kolmogorov Smirnov and Shapiro Wilk tests will be used to test the normal distribution of data. For comparing groups (POI/control) the student t-test will be used for variables that have a normal distribution, and the Mann Whitney U test will be used for variables that have not a normal distribution. The ROC analysis will be applied for the determination of cut-off point for variables. Moreover, Spearman correlation test will be used for the relationship of between variables. SPSS for Windows 22.0 and Medcalc programs will be used for statistical analysis. p<0.05 will be accepted as statistical significance.

#### 3. Outcome Measures

Primary Outcome Measures: Soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin concentrations

#### 4. Endpoints of the study:

The primary outcome in these analyses will compare serum soluble fms-like tyrosine kinase-1, proangiogenic protein placental growth factor, and niacin levels in study group and control group.

#### 5. Limitations and strengths:

There will strengths of this study. The women participating in the study had idiopathic POI and had not received treatment.

#### 6. Certain Agreements

The authors declare that they have no conflict of interest.

#### 7. Results Point of Contact

**Corresponding Author:** Ali Ovayolu, Department of Obstetrics and Gynecology, Cengiz Gokcek Women's and Children's Hospital, Gaziantep, Turkey, drovayolu@yahoo.com

**Address:** Osmangazi Mahallesi, Cengiz Gokcek Kadın Hastaliklari ve Dogum Hastanesi, 27010 Gaziantep, Turkey

**GSM:** +90 (532) 640 40 60

**Tel.:** +90.342 360 08 88

**Fax:** +90.342 360 02 90